CLINICAL TRIAL: NCT06251557
Title: Additional Effects of Lumbopelvic Massage and Exercise Training to Standard Urotherapy and Biofeedback Therapy in Children With Lower Urinary Tract Dysfunction
Brief Title: Effects of Lumbopelvic Massage and Exercise Training in Children With Lower Urinary Tract Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-23059
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Children; Lumbopelvic massage therapy; Lumbopelvic exercise; Biofeedback therapy; Urotherapy
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Exercise; Electromyography; Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbopelvic Massage and Exercise Training in addition to Standard Urotherapy and Biofeedback Therapy (Experimental): Group 1 will receive lumbopelvic massage and exercise training in addition to standard urotherapy and pelvic floor EMG biofeedback therapy.
  Interventions: Other: Lumbopelvic Massage; Other: Exercise Training; Device: Pelvic Floor Electromyography (EMG) Biofeedback Therapy; Behavioral: Standard Urotherapy
- Standard Urotherapy and Biofeedback Therapy (Active Comparator): Group 2 will receive only standard urotherapy and pelvic floor EMG biofeedback therapy.
  Interventions: Device: Pelvic Floor Electromyography (EMG) Biofeedback Therapy; Behavioral: Standard Urotherapy

INTERVENTIONS:
Other: Lumbopelvic Massage — 10 minutes abdominal massage and 10 minutes lower back massage will be applied in each session. It will take 20 minutes in total.
  Arms: Lumbopelvic Massage and Exercise Training in addition to Standard Urotherapy and Biofeedback Therapy
Other: Exercise Training — Exercise training will last approximately 10 minutes in each session. In the exercise training, lumbopelvic stabilization exercises (bridge, cat-and-cow and squatting exercises) will be performed for 10 repetitions, lumbopelvic flexibility exercises (child position, happy baby position, adductor muscle stretching, psoas muscle stretching) will be performed for 20 seconds and 5 repetitions, and diaphragmatic breathing exercises will be performed for 5 repetitions in supine, side lying and sitting positions.
  Arms: Lumbopelvic Massage and Exercise Training in addition to Standard Urotherapy and Biofeedback Therapy
Device: Pelvic Floor Electromyography (EMG) Biofeedback Therapy — Biofeedback therapy will be applied for 20 minutes in each session. During the application, adhesive surface electrodes will be placed on the perineum at 4 o'clock and 8 o'clock for each child. Through these electrodes, the activity signals of the muscles in that area will be recorded superficially. By monitoring the regional muscle activity, feedback is provided to increase and/or decrease the activity according to the activity pattern. As a result, pelvic floor biofeedback therapy will teach the child the correct use of the pelvic floor muscles. During the session, pelvic floor awareness and relaxation exercises specific to the child will be practiced with visual animations.
Behavioral: Standard Urotherapy — The anatomy of the urinary system and related structures, the causes of voiding dysfunction and symptoms will be explained to the family and the child with visuals. A written form including timed voiding during the day, appropriate fluid intake, correct toilet posture, adequate and balanced nutrition will be given.

SUMMARY:
Lower urinary tract dysfunctions (LUTD) are common in the pediatric population and include symptoms related to functional disorders. LUTD limits children and their parents socially, physically, and financially; leads to secondary comorbidities in the long term and negatively affects quality of life. Therefore, effective treatment of LUTD is important. Treatment options in children with LUTD include standard urotherapy, physiotherapy and rehabilitation practices, pharmacologic approaches, and Botulinum toxin type A injections. Pharmacologic treatment and invasive approaches have high side effect rates and compliance problems; therefore, conservative treatment methods should be completed first. The literature focuses on standard urotherapy, pharmacologic approaches and biofeedback therapy. However, to the best of our knowledge, there is no study in this population that comprehensively addresses the anatomical structures closely related to the pelvic floor with a more holistic perspective beyond the standard patient education and pelvic floor. Therefore, The aim of our study is to demonstrate the additional effects of massage therapy and exercise training for the lumbopelvic area in children with LUTD compared to standard urotherapy and pelvic floor biofeedback therapy in a randomized controlled design.

DETAILED DESCRIPTION:
Pediatric lower urinary tract dysfunction (LUTD) is a common and multifactorial health problem. A holistic perspective is required in treatment. Therefore, the aim of our study is to demonstrate the additional effects of massage therapy and exercise training for the lumbopelvic area in children with LUTD compared to standard urotherapy and pelvic floor biofeedback therapy in a randomized controlled design. At the beginning of our study, sample size was estimated using the G Power 3.1.9.7 program. Estimating that a 30% difference between the two groups is clinically significant (80% improvement in the score in the research arm and 50% in the control arm), with 80% power and a margin of error of 0.05 in the one-way hypothesis design, the minimum number of samples that should be included in the study was determined for each A total of 62 volunteers were calculated for the group, 31 of which were volunteers. Anticipating a 10% loss rate in volunteers during the study period, the final sample size was calculated as 68 individuals in total, 34 individuals for each research arm. The study will include 68 volunteer children aged 7-15 years with symptoms associated with functional LUTD, accompanied by their parents. Children will be randomly assigned to 2 separate groups according to an online computer generated, gender stratified block randomization list. Group 1 will receive lumbopelvic massage and exercise training in addition to standard urotherapy and pelvic floor EMG biofeedback therapy. Group 2 will receive only standard urotherapy and pelvic floor EMG biofeedback therapy. The treatments will be applied 2 days a week for 6 weeks. Children will be evaluated at the beginning of the study and at the end of the treatment (6th week). The primary outcome measure is the "Dysfunctional Voiding and Incontinence Score". Secondary outcome measures are 3-day voiding and defecation diaries data, uroflowmetry parameters and residual urine volume after voiding by pelvic ultrasound. SPSS program will be used for data analysis. SPSS program will be used for data analysis. In the comparison of numerical data between 2 independent groups, "Independent Groups T Test" will be used when parametric assumptions are met and "Mann-Whitney U test" will be used when parametric assumptions are not met. In the analysis of change within the dependent group, "Significance Test of the Difference Between Two Pairs" will be used when parametric assumptions are met and "Wilcoxon Test" will be used when parametric assumptions are not met. In the examination of the change in outcome measurements over time, the effect of the treatments in both groups on the dependent variables in all evaluations (In-group factor, Time; pre-treatment and post-treatment) will be tested with "Repeated Measures of Anova" using Treatment Group*Time (2*2) factors. Type-1 error level for statistical significance will be based on 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7 and 15
* Presence of symptoms of functional lower urinary tract dysfunction
* Do not have a condition (such as autism, ADHD-Attention Deficit and Hyperactivity Disorder) that would prevent cooperation with the assessments and interventions in the study
* Consented to participate in the study by their parents

Exclusion Criteria:

* Symptomatic urinary tract infection,
* A neurological disease,
* Neurogenic bladder/bowel diagnosis,
* Monosymptomatic enuresis,
* Anatomical anomaly that may affect bladder/bowel function,
* Fecal incontinence,
* Disruption of skin integrity or open wound at the massage site and
* An orthopedic problem that would prevent them from performing the exercises in the study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Symptom score | Change in symptom score from baseline up to end of 6th week
  Dysfunctional Voiding and Incontinence Symptoms Score (DVISS) Questionnaire will be used to evaluate the symptom score.

SECONDARY OUTCOMES:
Frequency of voiding, incontinence and defecation | Change in frequency of voiding, incontinence and defecation from baseline up to end of 6th week
  3-day voiding and defecation diary will be used to evaluate the frequency of voiding, incontinence and defecation.
Uroflowmeter parameters | Change in uroflowmeter parameters from baseline up to end of 6th week
  Uroflowmeter test report will be used to evaluate the maximum and average voiding rate data.
Residual urine volume after voiding | Change in residual urine volume after voiding from baseline up to end of 6th week
  Pelvic ultrasound will be used to evaluate residual urine volume after voiding.

CONTACTS AND LOCATIONS:
Locations (1):
- Burcu Sert, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695
- [Background] Akbal C, Genc Y, Burgu B, Ozden E, Tekgul S. Dysfunctional voiding and incontinence scoring system: quantitative evaluation of incontinence symptoms in pediatric population. J Urol. 2005 Mar;173(3):969-73. doi: 10.1097/01.ju.0000152183.91888.f6. PMID 15711352
- [Background] Morgan KE, Leroy SV, Corbett ST, Shepard JA. Complementary and Integrative Management of Pediatric Lower Urinary Tract Dysfunction Implemented within an Interprofessional Clinic. Children (Basel). 2019 Jul 30;6(8):88. doi: 10.3390/children6080088. PMID 31366055